CLINICAL TRIAL: NCT00005605
Title: Does Tamoxifen Prevent the Skeletal and Cardiovascular Morbidity of Chemotherapy in Premenopausal Women?
Brief Title: Tamoxifen to Prevent Bone Loss and Heart Disease in Premenopausal Women Receiving Chemotherapy for Stage I or Stage II Breast Cancer
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Seema Khan, MD, Northwestern University
Other Study IDs: NU 95B2; NU-95B2; NCI-G00-1737
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: osteoporosis; stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Tamoxifen group
- Chemotherapy group

SUMMARY:
RATIONALE: Tamoxifen may be able to increase bone density and decrease cholesterol in women who are undergoing chemotherapy for breast cancer.

PURPOSE: Clinical trial to study the effectiveness of tamoxifen in preventing bone loss and heart disease caused by chemotherapy treatment in premenopausal women who have stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the bone density in the femoral neck and lumbar spine and cholesterol levels in premenopausal women with stage I or II breast cancer treated with adjuvant chemotherapy with or without tamoxifen.
* Collect information regarding breast cancer risk factors, treatment, pathology, diet, activity levels, weight, and smoking in these patients.

OUTLINE: Patients are stratified according to type of treatment (adjuvant chemotherapy plus tamoxifen vs adjuvant chemotherapy alone).

Patients receive adjuvant chemotherapy with or without oral tamoxifen at the discretion of the treating physician.

Prior to starting chemotherapy, patients undergo blood draw to measure baseline levels of follicle-stimulating hormone, estradiol, total cholesterol, high-density lipoproteins, and low-density lipoproteins. Patients undergo baseline bone densitometry of the femoral neck and lumbar spine to assess bone density prior to starting chemotherapy or within 30 days of the first drug treatment. Laboratory studies and bone densitometry are repeated at years 1 and 2. A comparison is made between the study findings at baseline and at years 1 and 2.

PROJECTED ACCRUAL: A total of 80 patients (40 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage I or II breast cancer
* Must be scheduled to receive adjuvant chemotherapy with or without tamoxifen
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 35 to 50

Sex:

* Female

Menopausal status:

* Premenopausal by follicle-stimulating hormone and estradiol levels

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* See Disease characteristics

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with stage I or II breast cancer currently undergoing treatment with either chemotherapy or tamoxifen.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2000-02; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema A. Khan, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States